CLINICAL TRIAL: NCT07023731
Title: A Phase 1/2 Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of ARV-806 in Participants With KRAS G12D Mutated Advanced Solid Tumors
Brief Title: A Study to Evaluate ARV-806 in Adults With Advanced Cancer That Has the KRAS G12D Mutation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Arvinas Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ARV-806-101; 2025-521062-10-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: KRAS G12D Mutation; Advanced Solid Cancer
Keywords: KRAS G12D Mutation; Advanced Solid Tumors; KRAS G12D Mutated Advanced Solid Tumors; KRAS G12D Mutated Pancreatic Ductal Adenocarcinoma; Pancreatic Cancer; PDAC; Non-Small Cell Lung Cancer; NSCLC; Colorectal Cancer; Colon Cancer; CRC; Appendiceal Carcinoma; Cholangiocarcinoma; Endometrial Cancer; Esophageal Adenocarcinoma; Gallbladder Cancer; Gastric Cancer; Melanoma; Ovarian Cancer; Small Bowel Adenocarcinoma; Thyroid Cancer; advanced cancer; KRAS; G12D mutation; Pancreas cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Colorectal Neoplasms; Colonic Neoplasms; Cholangiocarcinoma; Endometrial Neoplasms; Adenocarcinoma Of Esophagus; Gallbladder Neoplasms; Stomach Neoplasms; Melanoma; Ovarian Neoplasms; Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1/Part A (Dose Escalation) (Experimental): Participants will receive ARV-806 at the assigned doses and regimen (weekly or every 2 weeks).
  Interventions: Drug: ARV-806
- Phase 2/Part B (Dose Expansion) (Experimental): Participants will receive ARV-806 at one of up to 2 dose levels/regimens selected from Part A)
  Interventions: Drug: ARV-806

INTERVENTIONS:
Drug: ARV-806 — Intravenous infusion at assigned dose and dosing schedule

SUMMARY:
This is a study to evaluate the safety and potential anti-tumor activity of an investigational agent called ARV-806 in Adults with Advanced Cancer having a specific KRAS mutation. This is an open-label study which means that participants and study staff will know that all participants will receive ARV-806.

Researchers think that ARV-806 can work by breaking down a specific protein with a mutation that is present in some tumors, which might help prevent or slow tumors from growing. This will be the first time ARV-806 will be used in people. The investigational drug will be given through a vein. This is called intravenous (IV) infusion.

This study will include 2 parts.

In Part A (Phase 1), different small groups of participants will receive lower to higher doses of ARV-806. Adults with advanced cancers having a specific KRAS mutation will be included.

In Part B (Phase 2), participants will be assigned to receive one of up to 2 dose levels decided by the information from Part A. Part B will include participants with advanced pancreatic ductal cancer having a specific KRAS mutation.

ELIGIBILITY:
Inclusion Criteria:

Part A:

* Histological or cytological diagnosis of unresectable or metastatic solid tumor malignancy, AND
* Must have evidence of KRAS G12D mutation in tumor tissue or blood (circulating tumor deoxyribonucleic acid [ctDNA]), AND
* Must have received prior standard-of-care (SOC) therapy appropriate for their type and stage of disease and have no other available treatment options with curative intent, or, in the opinion of the investigator, would be unlikely to tolerate or derive clinically meaningful benefit from appropriate SOC therapy, AND
* Must have at least 1 measurable lesion

Part B:

* Histological or cytological diagnosis of unresectable or metastatic pancreatic ductal adenocarcinoma (PDAC) with KRAS G12D mutation status confirmed by local testing of tumor tissue using a validated molecular or next-generation sequencing (NGS) testing, AND
* Must be willing to provide archival tumor tissue or willing to undergo pretreatment biopsy, AND
* Must have received at least one prior standard of care systemic therapy for PDAC (systemic therapy received in the neoadjuvant or adjuvant setting is allowed), AND
* Participants must have at least 1 measurable lesion

Part A / Part B:

* Eastern Cooperative Oncology Group performance status of 0 or 1,
* Participants with adequate organ function,
* Participants must accept and follow pregnancy prevention guidance.

Exclusion Criteria:

Part A / Part B:

* Active brain metastases
* Carcinomatous meningitis
* Uncontrolled hypertension despite optimal medical therapy
* Prior treatment with a KRAS G12D or a KRAS G12C targeting therapy (pan-KRAS inhibitor/degrader included)
* Participants with an inability to comply with listed prohibited treatments
* Systemic anticancer therapy within 2 weeks or 5 half-lives (whichever is shorter) or radiation therapy (excluding palliative radiation) within 2 weeks prior to the study intervention treatment. If the last immediate anticancer treatment contained an antibody-based agent(s), then an interval of 28 days or 5 half-lives (whichever is shorter) of the agent(s) is required prior to receiving the study intervention treatment.
* Standard 12-lead electrocardiogram that demonstrates clinically relevant abnormalities that may affect participant safety or interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2029-04-02 (Estimated)

PRIMARY OUTCOMES:
Part A (Phase 1): Number of dose-limiting toxicities of ARV-806 | 28 days from first ARV-806 administration
  Number of participants within a dose escalation cohort with adverse events (AEs) meeting protocol defined dose limiting toxicities during cycle 1 (28 days).
Part A (Phase 1): Number of participants with AEs | From the study baseline to at least 28 days after last dose of ARV-806
  AEs as characterized by type, frequency, severity (as graded by National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE]), timing, seriousness, and relationship to study intervention as a measure of safety and tolerability
Part B (Phase 2): Overall Response Rate (ORR) | Approximately 2 years
  ORR is a parameter measuring the anti-tumor activity of ARV-806. ORR is the percentage of participants for whom the study treatment resulted in a complete response or partial response of the disease under study. It is measured using CT/MRI and RECIST 1.1 criteria per investigator assessment.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ARV-806 (Part A): Area under the plasma or blood concentration-time profile during a dosing interval (AUC0-tau) | At predefined intervals throughout the treatment period, up to approximately 6 months after first dose of ARV-806.
PK of ARV-806 (Part A): Area under the plasma or blood concentration time profile from time zero to the time of the last quantifiable concentration (Clast) (AUC0-last) | At predefined intervals throughout the treatment period, up to approximately 6 months after first dose of ARV-806
PK of ARV-806 (Part A): Maximum plasma or blood concentration (Cmax) | At predefined intervals throughout the treatment period, up to approximately 6 months after first dose of ARV-806.
PK of ARV-806 (Part A): Minimum observed concentration (Cmin) | Timeframe: At predefined intervals throughout the treatment period, up to approximately 6 months after first dose of ARV-806.
PK of ARV-806 (Part A): Plasma or blood clearance (CL) | At predefined intervals throughout the treatment period, up to approximately 6 months after first dose of ARV-806.
PK of ARV-806 (Part A): Time for Cmax (Tmax) | At predefined intervals throughout the treatment period, up to approximately 6 months after first dose of ARV-806.
PK of ARV-806 (Part A): Volume of distribution (Vd) | At predefined intervals throughout the treatment period, up to approximately 6 months after first dose of ARV-806
Part A: Overall Response Rate (ORR) | Approximately 2 years
Part A: Time to Response (TTR) | Approximately 2 years
Part A: Duration of Response (DOR) | Approximately 2 years
Part A: Disease Control Rate (DCR) | Approximately 2 years
Part B: Number of participants with AEs | From the study baseline to at least 28 days after last dose of ARV-806
Part B: ARV-806 whole blood pre-dose concentration | At predefined intervals throughout the treatment period, up to approximately 6 months after first dose of ARV-806
Part B: Time to Response (TTR) | Approximately 2 years
Part B: Duration of Response (DOR) | Approximately 2 years
Part B: Disease Control Rate (DCR) | Approximately 2 years

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Clinical Trial Site, Grand Rapids, Michigan
  - Clinical Trial Site, Huntersville, North Carolina
  - Clinical Trial Site, San Antonio, Texas
  - Clinical Trial Site, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No